CLINICAL TRIAL: NCT01895556
Title: A Study of the Effect of Information About the Relationship Between HIV Transmission and Circumcision on Subsequent Sexual Behavior, and the Demand for Circumcision Among Circumcised and Uncircumcised Men in Malawi, Africa.
Brief Title: Information About HIV Transmission and Circumcision on Subsequent Sexual Behavior, and the Demand for Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca Thornton (Other)
Responsible Party: Sponsor-Investigator, Rebecca Thornton, Assistant Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FSG09-Thornton
Record Dates: First submitted 2013-06-28; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Sexual Behavior; Dis-inhibition
Keywords: Malawi; Risk Compensation; Male Circumcision; Demand
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Information (Experimental): Information about male circumcision and HIV risk
  Interventions: Other: Information
- Control (Placebo Comparator): Control
  Interventions: Other: Control

INTERVENTIONS:
Other: Information
  Arms: Information
Other: Control
  Arms: Control

SUMMARY:
The purpose of this study is to measure the behavioral effects of learning information about male circumcision and HIV risk on sexual behavior and the demand for male circumcision.

ELIGIBILITY:
Inclusion Criteria:

* The study will involve men between the ages of 25 and 40

Exclusion Criteria:

* None

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Condom use | One year after baseline survey
  frequency of reported condom use across all sexual acts (never, sometimes, always)

SECONDARY OUTCOMES:
Male circumcision | One year after baseline survey
  Circumcision, willingness to circumcise, circumcision of son
Condom purchases | one year after baseline survey
  number of condoms purchased
number of sexual partners | one year after baseline survey
  number of partners over last year with which individual has engaged in vaginal, anal, oral intercourse

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Thornton, PhD, Principal Investigator — University of Michigan; Susan Godlonton, PhD, Study Director — University of Michigan